CLINICAL TRIAL: NCT03034928
Title: Clinical Biocompatibility Evaluation of Contact Lens Coatings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-E002
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2020-02-18 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Refractive Errors; Ametropia
MeSH Terms: conditions — Refractive Errors | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Test 1/Control 1, then Control 2/Test 2 (Other): Contact lens with investigational coating 1 in right eye, with balafilcon A contact lens in left eye during Period 1, followed by balafilcon A contact lens in right eye, with contact lens with investigational coating 2 in left eye during Period 2. Each lens pair worn contralaterally for approximately 2 hours, with 2 to 8 days between pairs.
  Interventions: Device: Contact lens with investigational coating 1; Device: Balafilcon A contact lens; Device: OPTI-FREE® RepleniSH® MPDS; Device: Contact lens with investigational coating 2
- Test 2/Control 2, then Control 1/Test 1 (Other): Contact lens with investigational coating 2 in right eye, with balafilcon A contact lens in left eye during Period 1, followed by balafilcon A contact lens in right eye, with contact lens with investigational coating 1 in left eye during Period 2. Each lens pair worn contralaterally for approximately 2 hours, with 2 to 8 days between pairs.
  Interventions: Device: Contact lens with investigational coating 1; Device: Balafilcon A contact lens; Device: OPTI-FREE® RepleniSH® MPDS; Device: Contact lens with investigational coating 2
- Control 1/Test 1, then Test 2/Control 2 (Other): Balafilcon A contact lens in right eye, with contact lens with investigational coating 1 in left eye during Period 1, followed by contact lens with investigational coating 2 in right eye, with balafilcon A contact lens in left eye during Period 2. Each lens pair worn contralaterally for approximately 2 hours, with 2 to 8 days between pairs.
  Interventions: Device: Contact lens with investigational coating 1; Device: Balafilcon A contact lens; Device: OPTI-FREE® RepleniSH® MPDS; Device: Contact lens with investigational coating 2
- Control 2/Test 2, then Test 1/Control 1 (Other): Balafilcon A contact lens in right eye, with contact lens with investigational coating 2 in left eye during Period 1, followed by contact lens with investigational coating 1 in right eye, with balafilcon A contact lens in left eye during Period 2. Each lens pair worn contralaterally for approximately 2 hours, with 2 to 8 days between pairs.
  Interventions: Device: Contact lens with investigational coating 1; Device: Balafilcon A contact lens; Device: OPTI-FREE® RepleniSH® MPDS; Device: Contact lens with investigational coating 2

INTERVENTIONS:
Device: Contact lens with investigational coating 1 — Contact lens with investigational coating 1 pre-cycled in OPTI-FREE® RepleniSH® Multi-Purpose Disinfecting Solution (MPDS)
  Other Names: Test 1
Device: Balafilcon A contact lens — Balafilcon A contact lens pre-cycled OPTI-FREE® RepleniSH® MPDS
  Other Names: Bausch & Lomb PureVision™; Control 1; Control 2
Device: OPTI-FREE® RepleniSH® MPDS — Multipurpose contact lens solution
Device: Contact lens with investigational coating 2 — Contact lens with investigational coating 2 pre-cycled in OPTI-FREE® RepleniSH® MPDS
  Other Names: Test 2

SUMMARY:
The primary objective is to evaluate corneal staining observed after 2 hours of wear with contact lenses with investigational coating against PureVision™ lenses, all pre-cycled with OPTI-FREE® RepleniSH® multi-purpose disinfection solution.

DETAILED DESCRIPTION:
In this contralateral crossover study, qualifying subjects will wear a total of 2 pairs of study contact lenses. Lenses will be worn according to a randomized lens sequence assignment. Each pair will consist of a test lens (Test 1 or Test 2) and a control lens.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and must sign an Informed Consent;
* Successful wearer of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Manifest cylinder less than or equal to 1.50 diopter (D) in each eye;
* Best Corrected Visual Acuity (BCVA) 20/25 or better in each eye;
* VA with habitual spectacles 20/40 in both eyes (OU) or better and willing to wear spectacles as needed during the washout period and during study lens exposure;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any anterior segment infection, inflammation, abnormality or disease that contraindicates contact lens wear;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated;
* History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye;
* Ocular or intra-ocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study;
* Current or history of pathologically dry eye in either eye that would preclude contact lens wear;
* Current or history of herpetic keratitis in either eye;
* Eye injury in either eye within 12 weeks immediately prior to enrollment;
* History of intolerance or hypersensitivity to any component of the study lenses or solutions;
* Habitual contact lenses worn in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment;
* Use of topical ocular medications and artificial tear or rewetting drops that would require instillation during contact lens wear;
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Manager, Trial Management Operations, Study Director — Alcon, A Novartis Division
Locations (1):
- Alcon Investigative Site, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 1 study center located in the United States (US).
Pre-assignment Details: All 33 subjects enrolled were randomized. This reporting group includes all randomized subjects (33).
Period: Period 1, First 2 Hours of Wear
Arm/Group | Test 1/Control 1, Then Control 2/Test 2 | Test 2/Control 2, Then Control 1/Test 1 | Control 1/Test 1, Then Test 2/Control 2 | Control 2/Test 2, Then Test 1/Control 1
Started (Started = Randomized) | 8 | 8 | 9 | 8
Completed | 8 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period Between Lens Wear
Arm/Group | Test 1/Control 1, Then Control 2/Test 2 | Test 2/Control 2, Then Control 1/Test 1 | Control 1/Test 1, Then Test 2/Control 2 | Control 2/Test 2, Then Test 1/Control 1
Started | 8 | 8 | 9 | 8
Completed | 8 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0
Period: Period 2, Second 2 Hours of Wear
Arm/Group | Test 1/Control 1, Then Control 2/Test 2 | Test 2/Control 2, Then Control 1/Test 1 | Control 1/Test 1, Then Test 2/Control 2 | Control 2/Test 2, Then Test 1/Control 1
Started | 8 | 8 | 9 | 8
Completed | 8 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects exposed to any study lens (Safety Analysis Set).
Groups:
- Overall: Contact lens with investigational coatings and balafilcon A contact lens worn contralaterally during Period 1 and Period 2.
Arm/Group | Overall
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 27
  Black or African American | 5
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Multi-Racial | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Area of Solution-related Corneal Staining
Description: Percent of solution-related corneal staining area was assessed first in each of the 5 corneal regions: central, superior, nasal, inferior, and temporal. The average of corneal staining area was then calculated as the average over all 5 regions. A higher percentage reflects more damage to the corneal surface. Both eyes contributed to the analysis. No hypotheses were formulated; no inferences were made and only descriptive statistics were used in the reporting.
Time Frame: Day 1 after 2 hours of wear, each product
Population: This analysis population includes all randomized subjects who satisfied protocol-specified criteria (Full Analysis Set).
Measure: Mean (Standard Deviation); unit: percentage of area
Groups:
- Test 1: Contact lens with investigational coating 1 worn for approximately 2 hours during Period 1 or Period 2
- Control 1: Balafilcon A contact lens worn contralaterally to Test 1 for approximately 2 hours during Period 1 or Period 2
- Test 2: Contact lens with investigational coating 2 worn for approximately 2 hours during Period 1 or Period 2
- Control 2: Balafilcon A contact lens worn contralaterally to Test 2 for approximately 2 hours during Period 1 or Period 2
Arm/Group | Test 1 | Control 1 | Test 2 | Control 2
Number analyzed (Participants) | 33 | 33 | 33 | 33
percentage of area | 7.01 (10.54) | 12.82 (17.93) | 13.54 (17.20) | 7.58 (10.34)

ADVERSE EVENTS:
Time Frame: Baseline through study completion, approximately 8 days
Description: An adverse event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, whether or not related to the investigational medical device. AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol. Safety Analysis Set, based on treatment-specific exposure.
Groups:
- Test 1: All subjects exposed to contact lens with investigational coating 1 during Period 1 or Period 2
- Test 2: All subjects exposed to contact lens with investigational coating 2 during Period 1 or Period 2
- Control: All subjects exposed to balafilcon A contact lens during Period 1 or Period 2
Arm/Group | Test 1 | Test 2 | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT03034928/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/28/NCT03034928/SAP_001.pdf